CLINICAL TRIAL: NCT00499928
Title: An Open-Label Study to Investigate the Excretion and Metabolic Disposition of a Single, Oral Dose of [14C]-SB-751689 (a Calcium-Sensing Receptor Antagonist) in Healthy Male Subjects and Healthy Postmenopausal Female Subjects
Brief Title: A Study To Investigate The Metabolism And Excretion Of 14C SB-751689 Given To Healthy Males And Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR9106327
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Osteoporosis
Keywords: SB-751689; osteoporosis; metabolism; excretion
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: SB-751689

SUMMARY:
This study will examine the biological fate of radioactive SB-751689 administered to healthy males and healthy postmenopausal women. Subjects will receive a single oral dose of radioactive SB-751689. Excreta and blood samples will be taken over the course of 7 days. This study will help determine the major route of elimination of SB-751689 in humans. It will also provide samples (blood, plasma, urine, and stools) for analysis of metabolites, if any.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males of age 35 to 65 years, inclusive, or healthy ambulatory postmenopausal women defined as being amenorrheic for at least 2 years and 40 to 65 years of age, inclusive, at screening with FSH levels consistent with menopause. Healthy postmenopausal women, who are between ages 40 to 50 years, inclusive, must also have a documented history of bilateral oophorectomy (with or without hysterectomy) and be at least 6 weeks post-surgery.)
* Non-smokers
* Body weight > or = 50 kg and BMI within the range 19 - 32 kg/m2
* A history of regular bowel movements
* Capable of giving written informed consent

Exclusion Criteria:

* Any clinically relevant biological or physical abnormality found or reported at screening which, in the opinion of the investigator, is clinically significant and would preclude safe participation in this study
* QTc interval of > 450 msec at screening
* Positive urine drug screen at screening
* Positive urine test for alcohol at pre-dose
* Positive for HIV at screening
* Chronic hepatitis B and C, as evidenced by positive Hepatitis B surface antigen or Hepatitis C antibody
* Urinary cotinine levels indicative of smoking at screening
* History of smoking or use of nicotine containing products within one year of the study or >10 pack-year history of smoking overall
* History of regular alcohol consumption exceeding 7 units/week for women and 14 units/week for men within 6 months of screening
* History of drug abuse within 6 months of the study
* Participation in a clinical study and received a drug or a new chemical entity with 30 days or 5 half-lives, or twice the duration of the biological effect of any drug prior to the first dose of the current study medication
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Subjects who have received a total body radiation dose of greater than 5.0 mSv or exposure to significant radiation in the 12 months prior to this study
* Radiation exposure from the previous 3 year period is over 10 mSv for subjects who have been exposed to ionizing radiation above background as a result of their work with radiation as category A workers or as a result of research studies they may have been involved in. Clinical exposure will not be included
* Condition that could interfere with the accurate assessment and recovery of radiocarbon [14C]
* Use of prescription or nonprescription drugs including antacids, including vitamins, herbal and dietary supplements within 7 days prior to the first dose of study medication.
* Consumption of red wine, grapefruit, grapefruit juice or grapefruit-containing products within 14 days prior to the first dose of study medication
* Donation of blood in excess of 500 mL within 56 days prior to dosing.
* Evidence of renal, hepatic or biliary impairment
* History of serious gastrointestinal disease or history of a gastrointestinal surgical procedure that might affect the absorption of SB-751689
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation
* History of clinically significant cardiovascular disease
* History of pernicious anemia, pancreatitis, osteosarcoma or kidney stones.
* Conditions that might alter bone metabolism, including hyperparathyroidism, hypoparathyroidism, hyperthyroidism, hypothyroidism, Paget's disease, myeloma, malabsorption, or Cushing's syndrome, and hypogonadism (for male subjects), hypocalcemia, hypercalcemia, hypophosphatemia, hypomagnesemia, hypermagnesemia, osteopetrosis, osteomalacia, and recent history of fracture or prolonged bed rest
* Liver function tests, PTH, or CPK outside the reference range at screening
* Males unwilling to refrain from fathering a child during the study and for 14 days after

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The total amount of administered radioactivity recovered in excreta and the primary route of excretion over 7 days | over 7 days

SECONDARY OUTCOMES:
The amount of radioactivity associated with blood vs. plasma. The total amount radioactivity vs. SB-751689 radioactivity (metabolite vs. parent) over 7 days | over 7 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, M.D., Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Madison, Wisconsin, United States